CLINICAL TRIAL: NCT02997839
Title: Sleep Disruption in Post-operative Patients in the Neurocritical Care Unit
Acronym: SDPPNCU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in design to observational study
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00092868
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Sleep Fragmentation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 2 (No Intervention): no intervention
- group 1 (Other): sleep disruption
  Interventions: Behavioral: sleep disruption

INTERVENTIONS:
Behavioral: sleep disruption — Group two will have interrupted sleep at time periods of 2 hours post operatively.
  Group two will be woken every 2 hours, which is the standard NCCU protocol.
  Other Names: group 2
  Arms: group 1

SUMMARY:
The role of sleep in patients admitted to the intensive care unit is an emerging field of research. There have been studies that show patients in the ICU have poor sleep including sleep fragmentation, multiple arousals, decreased stage 3 sleep and reduced REM sleep (1, 2, 3). Causes of poor sleep in the ICU include severity of illness, abnormal light exposure, and frequent arousals for medical care. Not only does poor sleep contribute to reduced cognitive function and delirium, but there are also implications for the immune system function and wound healing (4). Polysomnography is regarded as the gold standard for sleep studies, however it has limited utility in the ICU population (5) and alternative methods of sleep analysis need to be investigated to better understand the underlying physiologic mechanisms and subsequent cognitive effects.

DETAILED DESCRIPTION:
The importance of sleep for patients in the intensive care unit (ICU) has been well documented. Research has shown that the ICU has multiple risk factors for poor sleep, and that this has multiple effects on patient outcomes. Further research is needed to better define the best tool to use for measuring sleep stages in ICU patients. Furthermore, there is very limited data comparing sleep interruption in ICU patients and the effects on sleep architecture and cognition.

Hypothesis 1a: The number of episodes of rapid eye movements (REM), stage 1, stage 2, stage 3 sleep, sleep spindles, and alpha activity will increase while the total duration of activity and the duration of episodes will decline in the postoperative neurologic critical care unit (NCCU) with neurological checks every two hours over a 12 hour period of recording as compared to every 6 hours.

Hypothesis 1b: As the number of episodes of REM, stage 1, stage 2, stage 3 sleep, sleep spindles, and alpha activity increase while the total duration of activity and the duration of episodes decline in the postoperative NCCU with neurological checks every two hours over a 12 hour period of recording as compared to every 6 hours.

Hypothesis 2: The number of episodes, the total duration, and the interval durations, of REM, stage 1, stage 2, stage 3 sleep, sleep spindles, and alpha activity will be identical in the automated recordings as compared to human reading by a sleep trained Neurologist.

Hypothesis 3: The group with awakenings every two hours will report more objective sleepiness and perform psychomotor visual task (PVT) with increased time and reduced performance.

Performing this study will allow for validation of an automated EEG system for the interpretation of sleep. If this tool is a reliable method of sleep interpretation, it may be expanded to a larger population of ICU patients for further research on the effects of sleep deprivation. Additionally, it will add prospective data to the literature regarding the psychomotor effects of increased sleep interruption in ICU patients.

2. Objectives (include all primary and secondary objectives)

1. Detect the effects of disrupted sleep resulting from frequent neurological exams in the NCCU in post-surgical patients. The investigators will use an automated EEG detection system used in patients with continuous EEG (cEEG) monitoring to detect duration of sleep related EEG brain activity, number of intervals of activation, and the duration of the intervals for sleep activities including: REM, Stage 1, stage 2, and stage 3 sleep, sleep spindles, and alpha activity.
2. The investigators will study the precision, accuracy and bias of the automated algorithm by comparing it to the interpretations of two sleep trained neurologists who will read these recordings in a

   blinded manner independently of one another. The investigators will select records to validate the automatic scorer including the identification and duration of all aspects of the cEEG sleep recording during the first four hours of sleep recording for each patient. The investigators will compare the accuracy of identification and measured duration of REM, Stage one, stage two, stage 3 sleep, sleep spindles, and alpha activity.
3. Subjective measure of sleep assessment using the Richards-Campbell Sleep Questionnaire (RCSG).
4. Quantitative assessment of alertness using a psychomotor vigilance task (PVT).

ELIGIBILITY:
Inclusion Criteria:

* post operative back patients in the NCCU with no history of brain injury

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Detect the effects of disrupted sleep with quantitative EEG analysis | Up to 12 hours
  The investigators will use an automated EEG detection system used in patients with continuous EEG (cEEG) monitoring to detect duration of sleep related EEG brain activity, number of intervals of activation, and the duration of the intervals for sleep activities including: REM, Stage 1, stage 2, and stage 3 sleep, sleep spindles, and alpha activity.

SECONDARY OUTCOMES:
Precision, accuracy and bias of the automated cEEG algorithm by comparing it to the interpretations of sleep trained neurologists | Up to 4 hours
  Two sleep trained neurologists will read these recordings in a blinded manner independently of one another. The investigators will select records to validate the automatic scorer including the identification and duration of all aspects of the cEEG sleep recording during the first four hours of sleep recording for each patient. The investigators will compare the accuracy of identification and measured duration of REM, Stage one, stage two, stage 3 sleep, sleep spindles, and alpha activity.
Subjective measure of sleep assessment using the Richards-Campbell Sleep Questionnaire | Up to 12 hours
Quantitative assessment of alertness using a psychomotor vigilance task (PVT). | Up to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Nyquist, MD, Principal Investigator — Johns Hopkins school of medicine
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No